CLINICAL TRIAL: NCT00128947
Title: Pharmacokinetics of Mycophenolic Acid and Mycophenolate 7-O-Phenolic Glucuronide in Healthy Subjects With or Without Two Common Genetic Polymorphisms in the Promoter Region of Uridine Diphosphate Glucuronosyltransferase 1A9
Brief Title: Pharmacokinetics of Mycophenolate Mofetil in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050209; 05-CC-0209
Record Dates: First submitted 2005-08-09; First posted 2005-08-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-05

CONDITIONS: Healthy
Keywords: Immunosuppresant; Pharmacogenetics; Glucuronidation; Metabolism; UGT
MeSH Terms: interventions — Mycophenolic Acid

INTERVENTIONS:
Drug: Mycophenolic Acid
Drug: Mycophenolate 7-O-Phenolic Glucuronide

SUMMARY:
This study will examine how people differ in the way their bodies process and eliminate mycophenolate mofetil (MMF), a drug that is used to treat problems affecting the eye and immune system and to prevent organ rejection in transplant patients. MMF is metabolized by a group of enzymes called UGTs, each of which is made by a different gene. This study will investigate whether people with different UGT genes differ in how well their bodies use and remove MMF. The results may help scientists learn the best way to give MMF to patients.

Normal healthy volunteers between 18 and 55 years of age may be eligible for this study. Candidates are screened with a medical history, physical examination, and blood and urine tests, including a blood test for analysis of genes that control and regulate UGTs. Pregnant women and nursing mothers are excluded from the study. Women who are able to have a child and men who can father a child must either abstain from sex or use two reliable forms of birth control during the study and for 3 months after its completion.

Participants come to the NIH Clinical Center at 6:30 a.m. on the first day of the study and stay in the outpatient clinic for 12 hours. The next 4 mornings, they return to the Clinical Center for a single blood collection. The procedures for the 5 days are as follows:

Day 1

Upon arrival at the Clinical Center a catheter is inserted into the subject's arm vein. At 7:00 AM, the subject takes one dose of MMF by mouth with a glass of water. Small blood samples are collected through the catheter before the MMF dose and again at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours after taking the drug. Heart rate and blood pressure are measured before the blood collection and then every 4 hours. After the last blood sample is collected, the volunteer can return home.

Days 2-5

Volunteers come to the Clinical Center at 7:00 AM on study days 2, 3, 4, and 5 for a single blood draw, collected using a needle.

Volunteers are contacted by telephone 1, 2, and 3 months after completing the study to see how they are doing and to check on their pregnancy status and use of appropriate birth control.

DETAILED DESCRIPTION:
The immunosuppressant mycophenolate mofetil (MMF) is metabolized by several uridine diphosphate glucuronosyltransferases (UGTs), among which UGT1A9 is the most important enzyme. Two commonly occurring single nucleotide polymorphisms (SNPs) in the promoter region of the UGT1A9 gene have been shown to enhance UGT1A9 protein level and activity in vitro. This study is to investigate the potential in vivo effects of these two SNPs on the metabolism and hence the pharmacokinetics of MMF metabolites. One hundred and thirty healthy volunteers will be screened for the presence of UGT1A9 C-2152T and T-275A polymorphisms. Seventeen subjects who carry the variant alleles, along with 17 others who do not have the polymorphisms, will be selected to participate in the pharmacokinetic study. Pharmacokinetics of the metabolites mycophenolic acid (active) and mycophenolate 7-O-phenolic glucuronide (inactive) will be determined, and parameter values will be compared between the two groups. It is hypothesized that the metabolism of MMF is enhanced in subjects with the two SNPs, resulting in an increase in clearance and a decrease in the exposure of mycophenolic acid.

ELIGIBILITY:
INCLUSION CRITERIA:

* Normal healthy volunteers who are in good health as determined by medical history, physical examination, and baseline laboratory tests
* Age 18 - 55
* Both males and females
* Willingness to practice effective contraception during the study and for three months after the administration of MMF for women who are sexually active and have child bearing potential, and for sexually active males who have the potential to father a child. Barrier or non-hormonal methods will be allowed during the study, whereas the use of oral, injectable, or implantable hormones will be prohibited since drug interaction is known to occur between oral contraceptives and mycophenolate mofetil.
* Subjects who are able to understand and sign the informed consent form.

EXCLUSION CRITERIA:

* Children and adolescents less than 18 years of age
* Individuals who smoke or have excessive alcohol (greater than 1 beer or an equivalent alcoholic beverage per day)
* Pregnant women and nursing mothers
* Subjects with certain underlying diseases which include diabetes, cardiovascular diseases, liver diseases, cancer, and human immunodeficiency virus infection
* Individuals with compromised immune systems
* Subjects who have an active infection
* Individuals with history of biliary tract disease, and biliary or gastrointestinal surgery
* Subjects with persistent diarrhea or other gastrointestinal problems that could impede drug absorption
* Subjects with abnormal liver and kidney functions as determined by medication history and laboratory evaluation (AST and ALT less than or equal to 2 x upper normal limit, total bilirubin less than or equal to 1 mg/dL, serum creatinine less than or equal to 1.2 mg/dL, hemoglobin greater than or equal to 11 g/dL, WBC greater than or equal to 3.5 x 10(9)/L)
* Volunteers on chronic prescribed and over-the-counter medications, and dietary and herbal supplements within 4 weeks of study participation
* Subjects who are taking any medications that could potentially interact with MMF pharmacokinetically and pharmacodynamically such as eccinacea, iron preparations, antacids, bile-resin cholesterol lowering agents, and steroids.
* Volunteers with documented allergy to MMF
* Prior enrollment into a similar study within the past two months and enrollment in another study at the same time
* Subjects who are felt to be unwilling or unable to practice effective contraception methods or comply with protocol specifications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130
Dates: Start 2005-07; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Allison AC, Eugui EM. Mycophenolate mofetil and its mechanisms of action. Immunopharmacology. 2000 May;47(2-3):85-118. doi: 10.1016/s0162-3109(00)00188-0. PMID 10878285
- [Background] Bullingham R, Monroe S, Nicholls A, Hale M. Pharmacokinetics and bioavailability of mycophenolate mofetil in healthy subjects after single-dose oral and intravenous administration. J Clin Pharmacol. 1996 Apr;36(4):315-24. doi: 10.1002/j.1552-4604.1996.tb04207.x. PMID 8728345
- [Background] Srinivas TR, Kaplan B, Meier-Kriesche HU. Mycophenolate mofetil in solid-organ transplantation. Expert Opin Pharmacother. 2003 Dec;4(12):2325-45. doi: 10.1517/14656566.4.12.2325. PMID 14640931